CLINICAL TRIAL: NCT01224730
Title: A Food Effect and QTc Study of Perifosine in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 147
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2012-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perifosine 100 mg (Experimental): Perifosine 100 mg orally daily under Fed and Fasted conditions
  Interventions: Drug: perifosine

INTERVENTIONS:
Drug: perifosine — 100 mg daily
  Other Names: D-21266; KRX-0401

SUMMARY:
This is a Phase I study which will analyze any food-drug effects as well as QTc effects of perifosine. Safety and efficacy will also be evaluated.

Patients who complete the first 24 days on single agent perifosine may have the opportunity to 1) continue on single agent perifosine; 2) switch to the combination of capecitabine + perifosine; or 3) switch to the combination of sorafenib + perifosine.

DETAILED DESCRIPTION:
Exclusion Criteria:

1. Patients with prior exposure to perifosine.
2. Patients receiving any other chemotherapy, targeted agents, investigational agents or devices within four weeks (28 days) or 5 half-lives of the agent(s), whichever is longer, prior to Day1 of study treatment.
3. Patients must have finished radiotherapy 28 days prior to start of treatment. Radiotherapy is not permitted in the Treatment Phase. Palliative radiotherapy to single sites for symptom control is allowed only during the Continuation Phase. The clinical coordinator should be contacted prior to initiating radiotherapy in this setting.
4. Patients who have had a major surgical procedure, open biopsy, or significant traumatic injury ≤4 weeks prior to Day 1 of study treatment.
5. Patients with a serious non-healing wound, active ulcer, or untreated bone fracture.
6. Patients with known central nervous system (CNS) metastases. Patients with CNS metastases that have been treated and are stable and who do not require corticosteroid treatment for the metastases (off steroids > 4 weeks) will be allowed.
7. Serious active infection requiring parenteral antibiotics or antifungal therapy.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
9. Patients with known dipyrimidine dehydrogenase (DPD) deficiency or prior severe reaction to 5-FU (for patients electing to receive capecitabine therapy in the Continuation Phase).
10. Patients with known HIV or acute or chronic active Hepatitis B or Hepatitis C.
11. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would Limit compliance with study requirements.
12. Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), or New York Heart Association class II-IV congestive heart failure (Appendix B).
13. Female patients who are pregnant or lactating. All females of childbearing potential must have a negative serum pregnancy test within 72 hours of treatment. Women of childbearing potential and men with partners of child-bearing potential, must agree to employ adequate contraception to prevent pregnancy while on therapy and for 4 weeks after the completion of treatment (see Appendix C).
14. A history of additional risk factors for Torsades de Pointes (e.g. familial long QT syndrome, hypokalemia, heart failure (Appendix B), left ventricular hypertrophy, slow heart rate (<45 bpm)).
15. Required use of concomitant medications known to prolong the QT/QTc interval

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignancies
* Patients with adequate organ and marrow function

Exclusion Criteria:

* Patients previously treated with perifosine
* Patients receiving any other chemotherapy, targeted agents, investigational agents or devices within four weeks (28 days) prior to Day 1 of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2013-11-04 (Actual); Study Completion 2013-11-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of food on the PK profile and bioavailability of perifosine, and to evaluate the effects of perifosine treatment on ECG parameters | 24 days
  * To assess the Pharmacokinetic profile of perifosine when given to patients under fed and fasted conditions
  * To evaluate changes in other ECG parameters associated with perifosine treatment (ventricular rate, PR interval, QRS interval, QT interval)

SECONDARY OUTCOMES:
To evaluate the safety and efficacy of perifosine when given to patients with advanced malignancies | Up to 6 months
  * To evaluate the safety profile (adverse events) and efficacy (response rate, and time to progression) of all study patients treated with perifosine.
  * After Day 24, to evaluate the safety profile (adverse events) and efficacy (response rate and time to progression) of all study patients who remain on single agent perifosine, switch to the combination of capecitabine + perifosine or switch to the combination of sorafenib + perifosine.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Cullen, PhD, Study Director — Keryx / AOI Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Dallas, Texas
  - Houston, Texas